CLINICAL TRIAL: NCT03221036
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Examine the Efficacy and Safety of Intravenous Vedolizumab (300 mg) Infusion Treatment in Chinese Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Vedolizumab IV in Chinese Participants With Ulcerative Colitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-3033; U1111-1195-3994 (Other: World Health Organisation)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Moderately to Severely Active Ulcerative Colitis
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Induction Phase: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg intravenous (IV) infusion at Weeks 0, 2, and 6 during induction phase.
  Interventions: Drug: Vedolizumab IV
- Induction Phase: Placebo (Placebo Comparator): Matching placebo IV infusion at Weeks 0, 2, and 6 during induction phase.
  Interventions: Drug: Placebo
- Maintenance Phase: Vedolizumab 300 mg (Experimental): Participants who received vedolizumab IV 300 mg in induction phase and achieved clinical response at Week 10 will be randomized to receive vedolizumab 300 mg IV infusion at Weeks 14, 22, 30, 38, 46 and 54. Participants who did not achieve clinical response at Week 10 will receive vedolizumab 300 mg IV infusion every 4 weeks from Week 14 up to Week 58.
  Interventions: Drug: Vedolizumab IV
- Maintenance Phase: Placebo (Placebo Comparator): Participants who received vedolizumab IV 300 mg in induction phase and achieved clinical response at Week 10 will be randomized to receive placebo, IV infusion at Weeks 14, 22, 30, 38, 46 and 54. Participants who received matching placebo in the induction phase and achieved clinical response at Week 10 will continue to receive placebo at Week 14, 22, 30, 38, 46, and 54.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Arms: Induction Phase: Vedolizumab 300 mg; Maintenance Phase: Vedolizumab 300 mg
Drug: Placebo — Matching-placebo IV infusion
  Arms: Induction Phase: Placebo; Maintenance Phase: Placebo

SUMMARY:
The purpose of this study is to assess the effect of vedolizumab intravenous IV as induction and maintenance treatment in Chinese participants with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
The drug being tested in this study is called Vedolizumab. Vedolizumab will be administered as an intravenous (IV) infusion. This study will investigate the efficacy and safety of vedolizumab IV as induction and maintenance therapy in participants with moderately to severely active ulcerative colitis (UC).

The study will enroll approximately 302 moderately to severely active patients with ulcerative colitis.

The Induction Phase contained 2 cohorts of participants: Cohort 1 participants will be randomized 1:2 in a double-blinded manner to receive:

* Vedolizumab IV 300 mg
* Placebo IV

Cohort 2 participants will be treated with open-label vedolizumab. The second cohort was enrolled to ensure that the sample size of Induction Phase responders randomized into the Maintenance Study provided sufficient power for the Maintenance Study primary efficacy analysis.

Participants will receive induction therapy of Vedolizumab 300 mg or matching placebo, intravenous (IV) infusion at Weeks 0, 2, and 6. At Week 10, participants will be assessed for clinical response based on complete clinic Mayo score. Results of Week 10 clinical response will determine the treatment pathway in maintenance phase.

In the Maintenance Phase, participants who received vedolizumab in the induction phase and achieved clinical response at Week 10 will be randomized 1:1 in a double-blinded manner to receive vedolizumab IV 300 mg or placebo starting from Week 14 (i.e., Weeks 14, 22, 30, 38, 46, and 54).

This multi-center trial will be conducted in China. The overall time to participate in this study is 60 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone, 6 months after last dose of investigational product (IP) for a long term follow-up safety survey.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of ulcerative colitis (UC) established at least 3 months prior to Screening by clinical and endoscopic evidence corroborated by a histopathology report. Cases of UC established at least 6 months before randomization for which a histopathology report is not available will be considered based on the weight of evidence supporting the diagnosis and excluding other potential diagnoses and must be discussed with the sponsor on a case-by case basis before randomization.
2. Has moderately to severely active UC as determined by a complete Mayo score of 6-12 with an endoscopic subscore ≥2 within 10 days prior to the first dose of IP. The endoscopy can be performed during the Screening Phase (Day -10 to Day -5 to allow for central reading prior to first dose at Week 0).
3. Has evidence of UC extending proximal to the rectum (≥15 cm of involved colon).
4. Participants with extensive colitis or pancolitis of >8 years duration or left-sided colitis >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months of the initial Screening Visit (may be performed during screening).
5. Participants with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factors must be up-to-date on colorectal cancer surveillance (may be performed during screening).
6. Has demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents: corticosteroids, immunomodulators, or tumor necrosis factor alpha (TNF-α) antagonists.

Exclusion Criteria:

1. Has evidence of abdominal abscess or toxic megacolon at the initial Screening Visit.
2. Has had extensive colonic resection, subtotal or total colectomy.
3. Has an existing ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine. A history of ileostomy or colostomy that has been reversed may be acceptable.
4. Has had any previous exposure to approved or investigational anti-integrins (for example, natalizumab, efalizumab, etrolizumab, or AMG-181) or mucosal address in cell adhesion molecule-1 (MAdCAM-1) antagonist, or rituximab.
5. Has used a topical (rectal) treatment with 5-acetyl salicylic acid (5-ASA) or corticosteroid enemas/suppositories or traditional Chinese medications for treatment of UC within 2 weeks of the administration of the first dose of IP.
6. Currently requires or is anticipated to require surgical intervention for UC during the study.
7. Has a history or evidence of adenomatous colonic polyps that have not been removed or has a history or evidence of colonic mucosal dysplasia including low or high-grade dysplasia, as well as indeterminate for dysplasia.
8. Has a suspected or confirmed diagnosis of Crohn's enterocolitis, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
9. Has evidence of or has had treatment for C. difficile infection or other intestinal pathogen within 28 days prior to randomization.
10. Has chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection.
11. Has active or latent TB.
12. Has any identified congenital or acquired immunodeficiency (for example, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
13. Has any history of malignancy, except for the following: (a) adequately treated non-metastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to randomization; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to randomization. Subjects with remote history of malignancy (for example, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to randomization.
14. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
15. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist at Screening or prior to the administration of the first dose of IP at Week 0.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2027-09-24 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Induction Phase: Percentage of Participants with Clinical Response at Week 10 | Week 10
  Clinical response is defined as ≥3 points reduction in complete Mayo clinical score and ≥30% decrease from baseline score accompanied with ≥1 point decrease in rectal bleeding subscore or absolute rectal bleeding subscore ≤1. Mayo clinical score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0= normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.
Maintenance Phase: Percentage of Participants with Clinical Remission at Week 60 | Week 60
  Clinical remission is defined as complete Mayo clinic score ≤2 with no subscore >1. Mayo clinic score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Induction Phase: Percentage of Participants with Clinical Remission at Week 10 | Week 10
  Clinical remission is defined as complete Mayo clinic score ≤2 with no subscore >1. Mayo clinic score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.
Induction and Maintenance Phase: Percentage of Participants with Mucosal Healing at Weeks 10 and 60 | Weeks 10 and 60
  Mucosal healing is defined as Mayo endoscopic subscore ≤1. Mayo clinic score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.
Maintenance Phase: Percentage of Participants with Durable Clinical Response at Weeks 10 and 60 | Weeks 10 and 60
  Clinical response is defined as ≥3 points reduction in complete Mayo clinical score and ≥30% decrease from baseline score accompanied with ≥1 point decrease in rectal bleeding subscore or absolute rectal bleeding subscore ≤1. Mayo clinic score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.
Maintenance Phase: Percentage of Participants with Durable Clinical Remission at Weeks 10 and 60 | Weeks 10 and 60
  Clinical remission is defined as complete Mayo clinic score ≤2 with no subscore >1. Mayo clinic score is used to assess ulcerative colitis disease activity. It consists of 4 subscales: stool frequency, rectal bleeding, findings on endoscopy and physician's global assessment. Each subscale is scored on a scale of 0 to 3, where 0 = normal condition and 3 = severe disease condition. The total Mayo clinic score ranges from 0 to 12, with higher scores indicating more severe disease.
Maintenance Phase: Percentage of Participants Using Oral Corticosteroids at Baseline who have Discontinued Corticosteroids and are in Clinical Remission at Week 60 | Week 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (35):
- China (35):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanchang University, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Army Medical University, PLA, Chongqing, Chongqing Municipality
  - Army Specialty Medical Center of The Chinese People's Liberation Army, Chongqing, Chongqing Municipality
  - The 900th Hospital of The Chinese People's Liberation Army Joint Logistics Support Force, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Nanchang University, Shanghai, Shanghai Municipality
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b603b4db2bf003ab4a329?idFilter=%5B%22Vedolizumab-3033%22%5D